CLINICAL TRIAL: NCT04081701
Title: 68Ga(Gallium)-DOTATATE Positron Emission Tomography (PET)/MRI in the Diagnosis and Management of Somatostatin Receptor Positive Central Nervous System CNS Tumors.
Brief Title: 68-Ga DOTATATE PET/MRI in the Diagnosis and Management of Somatostatin Receptor Positive CNS Tumors.
Acronym: DOMINO-START
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1807019445
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: CNS Tumors; Meningioma; Esthesioneuroblastoma; Hemangioblastoma; Medulloblastoma; Paraganglioma; Pituitary Adenoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningioma; Esthesioneuroblastoma, Olfactory; Hemangioblastoma; Medulloblastoma; Paraganglioma; Pituitary Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meningioma (Other): Cohort of 30 subjects with meningioma.
  Interventions: Diagnostic Test: Ga68-DOTATATE-PET/MRI
- Non-Meningioma (Other): Cohort of 60 subjects with non-meningioma:
  (esthesioneuroblastoma, hemangioblastoma, medulloblastoma, paraganglioma, pituitary adenoma and SSTR-positive tumors metastatic to the brain)
  Interventions: Diagnostic Test: Ga68-DOTATATE-PET/MRI

INTERVENTIONS:
Diagnostic Test: Ga68-DOTATATE-PET/MRI — In patients with meningioma who are undergoing surgical planning, subjects will undergo a PET scan at the time of their pretreatment or preoperative standard of care MRI exam, prior to surgery performed for research purposes. Instead of the standard of care MRI exam, subjects will undergo a dedicated hybrid Gallium-68-DOTATATE PET/MRI.There will be up to two follow-up with Ga68-DOTATATE PET/MRI scans performed as standard of care.
  In patients with SSTR-positive CNS tumors that are non-meningioma, MRI is often performed to assess extent of disease. Subjects may be asked to undergo a PET scan for research purposes at the time of their standard of care MRI. Instead of the standard of care MRI exam, they may be asked to undergo a dedicated hybrid Gallium-68-DOTATATE PET/MRI.

SUMMARY:
The study population consists of patients who undergo resection for somatostatin receptor-positive (SSTR-positive) CNS tumors, focusing on meningioma, and including esthesioneuroblastoma, hemangioblastoma, medulloblastoma, paraganglioma, pituitary adenoma, and SSTR-positive systemic cancers metastatic to the brain, such as small cell carcinoma of the lung. The study indication is to determine the diagnostic utility of 68Ga-DOTATATE PET/MRI in the diagnosis and management of patients with SSTR-positive CNS tumors, specifically whether 68Ga-DOTATATE PET/MRI demonstrates utility distinguishing between tumor recurrence and post-treatment change. To date, the utility of Ga-68-DOTATATE PET/MRI in meningioma has not been explored. Investigators have over the past 3 months been able to accrue the largest case series of presently 12 patients in whom Ga-68-DOTATATE PET/MRI demonstrated utility in the assessment of meningioma, including assessment for postsurgical/postradiation recurrence, detection of additional lesions not visualized on MRI alone, and evaluation of osseous invasion. Based on this initial experience, investigators intend to study the impact of Ga-68-DOTATATE PET/MRI in the assessment of the extent of residual tumor in patients status post meningioma resection, specifically in patients in whom tumor location limits resectability, patients with World Health Organization (WHO) grade II/III disease, and patients with history of stereotactic radiosurgery (SRS) who develop postradiation change.

DETAILED DESCRIPTION:
Prior to the onset of this study, the utility of Ga-68-DOTATATE PET/MRI in meningioma had not been explored. The investigator's pilot study serving as the basis for the proposed protocol resulted in the - to the investigators' knowledge - largest case series of 21 patients in whom Ga-68 DOTATATE PET/MRI demonstrated utility in the assessment of meningioma, including assessment for postsurgical/postradiation recurrence, detection of additional lesions not visualized on MRI alone, and evaluation of osseous invasion. Based on this initial experience, investigators continued to study the impact of Ga-68-DOTATATE PET/MRI in the assessment of the extent of residual tumor in patients status post meningioma resection, specifically in patients in whom tumor location limits resectability, patients with WHO grade II/III disease, and patients with history of SRS who develop postradiation change.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of meningioma based on pathology reports and suspected recurrence or residual disease based on standard-of-care MRI
* Additionally, patients with other somatostatin receptor 2 positive brain tumors, including esthesioneuroblastoma, hemangioblastoma, medulloblastoma, paraganglioma, pituitary adenoma, and SSTR-positive systemic cancers metastatic to the brain will be considered for the purposes of obtaining feasibility data
* As the investigator's institution, PET/MRI scanner utilizes a 3 Tesla (T) magnet, patients who may be ineligible to undergo 3T MRI but may undergo 1.5 Tesla (T) MRI, will undergo a 1.5T MRI as per clinical standard-of-care and a Ga68-DOTATATE PET/CT with the PET portion to be fused with the 1.5T MRI utilizing fusion software.

Exclusion Criteria:

* Contraindications to gadolinium-based contrast agent
* History of allergic reaction to Gallium-68-DOTATATE
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether Ga-68-DOTATATE PET/MRI provides additional clinical benefit | Longitudinal assessment up to 10 years
  Diagnostic accuracy of Ga-68-DOTATATE PET/MRI will be compared to MRI alone. Correlative analyses will be performed including logistic regression/ Spearman correlation for continuous variables, and Mann-Whitney U tests for not normally distributed subgroups for variables allowing for dichotomization.

SECONDARY OUTCOMES:
Correlate Ga-68-DOTATATE PET/MR findings with histopathologic biomarker, SSTR2 expression | Longitudinal assessment up to 10 years
  Histopathologic biomarkers, including SSTR2 expression will be assessed for patients with meningioma, who undergo resection. Correlative analyses will be performed including logistic regression/ Spearman correlation for continuous variables, and Mann-Whitney U tests for not normally distributed subgroups for variables allowing for dichotomization.
Correlate Ga-68-DOTATATE PET/Magnetic Resonance(MR) findings with histopathologic biomarker, Ki67 | Longitudinal assessment up to 10 years
  Histopathologic biomarkers, including Ki67 will be assessed for patients with meningioma, who undergo resection. Correlative analyses will be performed including logistic regression/ Spearman correlation for continuous variables, and Mann-Whitney U tests for not normally distributed subgroups for variables allowing for dichotomization.
Correlate Ga-68-DOTATATE PET/MR findings with histopathologic biomarker, progesterone receptor | Longitudinal assessment up to 10 years
  Histopathologic biomarkers, including progesterone receptor will be assessed for patients with meningioma, who undergo resection. Correlative analyses will be performed including logistic regression/ Spearman correlation for continuous variables, and Mann-Whitney U tests for not normally distributed subgroups for variables allowing for dichotomization.
Correlate Ga-68-DOTATATE PET/MR findings with histopathologic biomarker, epidermal growth factor receptor (EGFR) | Longitudinal assessment up to 10 years
  Histopathologic biomarkers, including EGFR will be assessed for patients with meningioma, who undergo resection. Correlative analyses will be performed including logistic regression/ Spearman correlation for continuous variables, and Mann-Whitney U tests for not normally distributed subgroups for variables allowing for dichotomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Ivanidze, MD/Ph.D, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ivanidze J, Chang SJ, Haghdel A, Kim JT, Roy Choudhury A, Wu A, Ramakrishna R, Schwartz TH, Cisse B, Stieg P, Muller L, Osborne JR, Magge RS, Karakatsanis NA, Roytman M, Lin E, Pannullo SC, Palmer JD, Knisely JPS. [Ga68] DOTATATE PET/MRI-guided radiosurgical treatment planning and response assessment in meningiomas. Neuro Oncol. 2024 Aug 5;26(8):1526-1535. doi: 10.1093/neuonc/noae067. PMID 38553990
- [Derived] Kim SH, Roytman M, Madera G, Magge RS, Liechty B, Ramakrishna R, Pannullo SC, Schwartz TH, Karakatsanis NA, Osborne JR, Lin E, Knisely JPS, Ivanidze J. Evaluating diagnostic accuracy and determining optimal diagnostic thresholds of different approaches to [68Ga]-DOTATATE PET/MRI analysis in patients with meningioma. Sci Rep. 2022 Jun 3;12(1):9256. doi: 10.1038/s41598-022-13467-9. PMID 35661809
- [Derived] Ivanidze J, Roytman M, Skafida M, Kim S, Glynn S, Osborne JR, Pannullo SC, Nehmeh S, Ramakrishna R, Schwartz TH, Knisely JPS, Lin E, Karakatsanis NA. Dynamic 68Ga-DOTATATE PET/MRI in the Diagnosis and Management of Intracranial Meningiomas. Radiol Imaging Cancer. 2022 Mar;4(2):e210067. doi: 10.1148/rycan.210067. PMID 35275019